CLINICAL TRIAL: NCT07340450
Title: Comparison of Oral vs Intravenous Iron Therapy for the Treatment of Postpartum Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahida Islam Medical Complex (Other)
Responsible Party: Principal Investigator, Sidra Jalil Khan, PGR obstetrics and Gynaecology, Shahida Islam Medical Complex
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIMC-postpartumanemia-2025
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Anaemia
MeSH Terms: interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Intravenous Iron Therapy (Experimental): Participants received intravenous iron therapy for the treatment of postpartum anemia
  Interventions: Drug: Ferric Carboxy Maltose
- Group B: Oral Iron Therapy (Experimental): Participants received oral iron therapy for the treatment of postpartum anemia.
  Interventions: Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: Ferric Carboxy Maltose — Participants received Intravenous iron i.e ferric carboxymaltose (≤1,000 mg) were given to patients in Group "A" either as a single dose or as two doses spaced three days apart in 100 milliliters of 0.9% normal saline during a half-hour period.
  Arms: Group A: Intravenous Iron Therapy
Drug: Ferrous Sulfate — Participants given tablet Ferrous sulfate, 325 mg orally three times a day.
  Arms: Group B: Oral Iron Therapy

SUMMARY:
Postpartum anemia is a common condition associated with adverse maternal outcomes. This study aimed to compare the effectiveness of oral iron therapy versus intravenous iron therapy in women with postpartum anemia.

DETAILED DESCRIPTION:
This randomized, open-label, parallel-group study was conducted at Shahida Islam Medical College and Hospital, Lodhran, Pakistan. Women diagnosed with postpartum anemia who fulfilled the eligibility criteria were randomly allocated using a lottery method to receive either intravenous iron (ferric carboxymaltose) or oral iron therapy (ferrous sulfate). The primary outcome was the change in hemoglobin level from baseline to 6 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. All women with postpartum anaemia as per operational definition i.e Haemoglobin <11 g/dl at 24 hours after delivery (either caesarean or SVD).
2. Age 20-40 years.
3. BMI 19-25.
4. Pre-operative haemoglobin >10 g/dl.
5. Both primiparous and multiparous.
6. Both primigravida and multigravida.

   -

Exclusion Criteria:

1. Iron Intolerance or previous history of allergy to iron
2. Parenteral Iron hypersensitivity
3. Patients with thalassemia
4. Indication of blood transfusion
5. Patients with bleeding/ clotting disorders
6. Patients with postpartum haemorrhage
7. Patients with chronic diseases.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 122 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin level | Baseline to 6 weeks postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Shahida Islam Medical College and Hospital, Lodhran, Lodhrān, Punjab Province, Pakistan